CLINICAL TRIAL: NCT00743522
Title: Programming Implantable Cardioverter Defibrillators (ICDs) in Patients With Primary Prevention Indication to Prolong Time to First Shock
Brief Title: Programming Implantable Cardioverter Defibrillators in Patients With Primary Prevention Indication
Acronym: PROVIDE
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 448
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Shock
Keywords: Reducing shocks
MeSH Terms: conditions — Shock | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: PROVE Trial settings
  Interventions: Device: ICD/ CRT-D
- Experimental: Pre-selected settings
  Interventions: Device: ICD/ CRT-D

INTERVENTIONS:
Device: ICD/ CRT-D — Cardiac device

SUMMARY:
Although shock therapy is effective in terminating ventricular tachycardia (VT), it can be painful to the patient and repetitive shocks can decrease a patient's quality of life. Previous studies have suggested that one or more sets of aggressive device parameter settings may reduce the total number of shocks in primary prevention patients. In addition to shock therapies, antitachycardia pacing (ATP) is also available in ICDs to treat VT. The PROVIDE trial aims to prospectively study the effect of high detection rates, prolonged detection intervals, aggressive SVT discriminators, and extensive ATP therapy in prolonging the time to first shock in primary prevention patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary Prevention indication for ICD/ CRT-D

Exclusion Criteria:

* No prior documented history of spontaneous VT/VF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with approved ICD/CRT-D indications
Sampling Method: Probability Sample
Enrollment: 1670 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is the rate of first shock | Average follow-up period is 530 days
The primary safety endpoint of this study is the rate of arrhythmic syncope | Average follow-up period is 530 days

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Saeed, MD, Principal Investigator — Hall-Garcia Cardiology Associates
Locations (1):
- Hall-Garcia Cardiology Associates, Houston, Texas, United States

REFERENCES:
- [Result] Saeed M, Hanna I, Robotis D, Styperek R, Polosajian L, Khan A, Alonso J, Nabutovsky Y, Neason C. Programming implantable cardioverter-defibrillators in patients with primary prevention indication to prolong time to first shock: results from the PROVIDE study. J Cardiovasc Electrophysiol. 2014 Jan;25(1):52-9. doi: 10.1111/jce.12273. Epub 2013 Sep 24. PMID 24112717
- [Derived] Sanders P, Connolly AT, Nabutovsky Y, Fischer A, Saeed M. Increased Hospitalizations and Overall Healthcare Utilization in Patients Receiving Implantable Cardioverter-Defibrillator Shocks Compared With Antitachycardia Pacing. JACC Clin Electrophysiol. 2018 Feb;4(2):243-253. doi: 10.1016/j.jacep.2017.09.004. Epub 2017 Nov 15. PMID 29749945